CLINICAL TRIAL: NCT06911463
Title: Conscious Sedation With Suprainguinal Facia Iliaca Block Versus Ilioinguinal Iliohypogastric Block for Transcatheter Aortic Valve Implantation (TAVI)
Brief Title: Conscious Sedation With Suprainguinal Facia Iliaca Block Versus Ilioinguinal Iliohypogastric Block for TAVI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohammed Shabayek, Lecturer of Anesthesia, ICU and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: FMASU R30/2024/2025
Record Dates: First submitted 2025-03-22; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (F) (Active Comparator): suprainguinal fascia iliaca block group (SIFIB)
  Interventions: Other: suprainguinal fascia iliaca block group (SIFIB)
- Group II (I) (Active Comparator): iliohypogastric and ilioinguinal group (IL-IH)
  Interventions: Other: iliohypogastric and ilioinguinal group (IL-IH)
- Group III (C) (Other): control group patients received infiltration of 0.5% 10ml bupivacaine and 1% 10 ml lidocaine in the groin at the site of puncture
  Interventions: Other: Local infiltration

INTERVENTIONS:
Other: suprainguinal fascia iliaca block group (SIFIB) — The anterior superior iliac spine is identified by a high-frequency linear probe (SonoSite HFL50x, 15-6 MHz, 55-mm broadband linear array, USA) the inguinal ligament in the parasagittal plane, following appropriate disinfection and draping of the patient in the supine position. Then, the probe is moved medially, and the internal oblique muscle in the cranial direction, the sartorius muscle in the caudal direction, the bow-tie shape formed by these muscles, the underlying iliacus muscle, and the fascia iliaca surrounding it is visualized. (21) An 80-mm peripheral nerve block needle is inserted from the caudal side, and the iliac fascia is passed. After identification of the correct area following 2 to 3 mL of hydro-dissection, 40 mL of 0.25% bupivacaine is injected.
  Arms: Group I (F)
Other: iliohypogastric and ilioinguinal group (IL-IH) — Group II (I): iliohypogastric and ilioinguinal group (IL-IH) After preparation of the inguinal region sterile linear high frequency probe (SonoSite HFL50x, 15-6 MHz, 55-mm broadband linear array, USA) is placed between the iliac crest and costal margin (more cephalad than the usual location for ilioinguinal block). In this location, the ilioinguinal and iliohypogastric nerves in between the transverses abdominus and internal oblique are well defined (22) After visualization, a 22G 1.5-inch needle is used in out of-plane approach to reach the nerves. After identification of the correct area following 2 to 3 mL of hydro-dissection, 40 mL of 0.25% bupivacaine is injected (kayak sign).
  Arms: Group II (I)
Other: Local infiltration — patients receive infiltration of 0.5% 10ml bupivacaine and 1% 10 ml lidocaine in the groin at the site of puncture.
  Arms: Group III (C)

SUMMARY:
the aim of the present study is to compare suprainguinal fascia iliaca block and ilioinguinal-iliohypogastric (II-IH) nerve block in improving the quality of conscious sedation, including reducing patients' requirements for analgesia also better satisfaction for both patient and surgeon as regards patient outcome and decreasing the incidence of conversion to general anesthesia during TAVI procedure

ELIGIBILITY:
Inclusion Criteria:

* aged >20 years with severe aortic stenosis undergoing elective, non-emergent, non-urgent transfemoral Sapien 3TM (Edwards Lifesciences Corp., Irvine, CA, USA) or CoreValveTM (Medtronic, Minneapolis, MN, USA) implantation were included in the study

Exclusion Criteria:

* younger than 20 years

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the timing to the first rescue analgesia | Six months
  sedation score (RASS), and pain (numerical rating scale [NSR] from 0 [no pain] to 10 [unbearable pain]) at 0 time start of sedation and every 30 min till the end of the procedure then 1, 3, and 6 h after TAVI. While, Pain intensity was assessed using numeric rating scale (NRS 0-10; 0 = no pain; 10 = the worth pains imaginable) in five time-points intraoperatively (femoral artery cannulation (1), aortic valve system introduction (2), aortic valve system removal (3), vessel closure devices insertion (4), the end of the operation (5)). In addition, the need for post TAVI pacing, vascular complications at the TAVI access site during admission, and the length of hospital stay were recorded.
  Rescue analgesia will be given When NRS was more than 4, patient discomfort or doctor dis-satisfaction is detected, 0.5 mic /kg fentanyl will be given. The primary outcome is the timing to the first rescue analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No